CLINICAL TRIAL: NCT04423718
Title: Randomized, Double-Masked, Active-Controlled, Phase 3 Study of the Efficacy and Safety of High Dose Aflibercept in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Study of the Effects of High Dose Aflibercept Injected Into the Eye of Patients With an Age-related Disorder That Causes Loss of Vision Due to Growth of Abnormal Blood Vessels at the Back of the Eye
Acronym: PULSAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20968; 2019-003851-12 (EudraCT Number)
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Results first posted 2023-09-06 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: nAMD
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Up to Week 108: Participant and Investigator masked. Week 108 to Week 156: Participant and Investigator unmasked to treatment intervals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Aflibercept 2q8 (Active Comparator): In the double-masked study part (Years 1 and 2), Aflibercept 2 mg administered every 8 weeks after a loading phase. (Active Comparator) In Year 3, high dose aflibercept administered according to individual patient response. (Experimental)
  Interventions: Drug: Aflibercept High Dose VEGF Trap-Eye (BAY86-5321); Drug: Aflibercept VEGF Trap-Eye (Eylea, BAY86-5321)
- Aflibercept HDq12 (Experimental): Aflibercept high dose (HD) administered every 12 weeks after an initiation phase. Treatment intervals adjusted according to individual patient response.
  Interventions: Drug: Aflibercept High Dose VEGF Trap-Eye (BAY86-5321)
- Aflibercept HDq16 (Experimental): Aflibercept high dose administered every 16 weeks after an initiation phase. Treatment intervals adjusted according to individual patient response.
  Interventions: Drug: Aflibercept High Dose VEGF Trap-Eye (BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept High Dose VEGF Trap-Eye (BAY86-5321) — Solution in Vial, intravitreal (IVT) injection
Drug: Aflibercept VEGF Trap-Eye (Eylea, BAY86-5321) — Solution in Vial, 2 mg, intravitreal (IVT) injection
  Arms: Aflibercept 2q8

SUMMARY:
In this study researchers want to learn more about changes in visual acuity (clarity of vision) with a high dose treatment with Aflibercept (Eylea) in patients suffering from neovascular age-related macular degeneration (nAMD). Neovascular AMD is an eye disease that causes blurred vision or a blind spot due to abnormal blood vessels that leak fluid or blood into the light sensitive lining inside the eye (retina). The fluid buildup causes the central part of the retina (macula) responsible for sharp, straight-ahead vision to swell and thicken (edema), which distorts vision.

ELIGIBILITY:
Inclusion Criteria:

* Active subfoveal CNV secondary to nAMD, including juxtafoveal lesions that affect the fovea as assessed in the study eye.
* Total area of CNV (including both classic and occult components) must comprise greater than 50% of the total lesion area in the study eye.
* BCVA ETDRS letter score of 78 to 24 (corresponding to a Snellen equivalent of approximately 20/32 to 20/320) in the study eye.
* Decrease in BCVA determined to be primarily the result of nAMD in the study eye.
* Presence of IRF and/or SRF affecting the central subfield of the study eye on OCT.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of highly effective contraception for those participating in clinical studies.
* Other protocol-specified inclusion criteria.

Additional inclusion criteria for Year 3:

* At least one BCVA value and one central subfield retinal thickness (CST) value from measurements at one of the following visits: Visit 24 (Week 84), Visit 25 (Week 88) or Visit 26 (Week 92).
* Participant is enrolled at a site that participates in the extension period.

Exclusion Criteria:

* Causes of CNV other than nAMD in the study eye.
* Scar, fibrosis, or atrophy involving the central subfield in the study eye.
* Presence of retinal pigment epithelial tears or rips involving the central subfield in the study eye.
* Uncontrolled glaucoma (defined as IOP >25 mmHg despite treatment with anti-glaucoma medication) in the study eye.
* History of idiopathic or autoimmune uveitis in the study eye.
* Myopia of a spherical equivalent of at least 8 diopters in the study eye prior to any refractive or cataract surgery.
* History or clinical evidence of diabetic retinopathy, diabetic macular edema, or any retinal vascular disease other than nAMD in either eye.
* Evidence of extraocular or periocular infection or inflammation (including infectious blepharitis, keratitis, scleritis, or conjunctivitis) in either eye at the time of screening/randomization.
* Uncontrolled blood pressure (defined as systolic >160 mmHg or diastolic >95 mmHg).
* Any prior or concomitant ocular (in the study eye) or systemic treatment (with an investigational or approved, anti-VEGF or other agent) or surgery for nAMD, except dietary supplements or vitamins.
* Other protocol-specified exclusion criteria

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1011 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2024-08-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (235):
- United States (57):
  - Arizona Retina & Vitreous Consultants - Central Phoenix Phoenix, Phoenix, Arizona
  - Retina Consultants of Orange County - Fullerton, Fullerton, California
  - Northern California Retina Vitreous Associates - Mountain View Office, Mountain View, California
  - Azul Vision Pasadena, Pasadena, California
  - Retina Consultants San Diego - Poway, Poway, California
  - Retina Consultants of Southern California, Redlands, California
  - Kaiser Permanente Riverside Medical Center - Cardiology, Riverside, California
  - Perlman Medical Offices at UC San Diego Health - Endocrinology, San Diego, California
  - Retina Consultants of Southern Colorado, PC, Colorado Springs, Colorado
  - New England Retina Associates, New London, Connecticut
  - Rand Eye Institute, Deerfield Beach, Florida
  - Retina Group of Florida - Fort Lauderdale, Fort Lauderdale, Florida
  - Vitreo Retinal Associates PA - The Millennium Center Location, Gainesville, Florida
  - Florida Retina Institute- Jacksonville Oak, Jacksonville, Florida
  - Florida Eye Associates - Melbourne Main Office, Melbourne, Florida
  - Retina Macula Specialists Of Miami - LeJeune Road Office, Miami, Florida
  - Florida Retina Institute - Orlando, Orlando, Florida
  - Retina Specialty Institute - Pensacola, Pensacola, Florida
  - Retina Vitreous Associates of Florida - Saint Petersburg, St. Petersburg, Florida
  - Southern Vitreoretinal Associates, P.L. - Tallahassee, Tallahassee, Florida
  - Retina Consultants of Hawaii - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Retina Associates IL, Elmhurst, Illinois
  - University Retina and Macula Associates, Oak Forest, Illinois
  - Wolfe Eye Clinic - Des Moines, West Des Moines, Iowa
  - The Retina Care Center - Baltimore, Baltimore, Maryland
  - Ophthalmic Consultants of Boston - Boston, Boston, Massachusetts
  - Vitreo Retinal Surgery PA - Edina, Edina, Minnesota
  - Retina Consultants of Nevada - Summerlin, Las Vegas, Nevada
  - Retina Center of New Jersey, Bloomfield, New Jersey
  - NJ Retina - Edison Office, Edison, New Jersey
  - Eye Associates of New Mexico - Albuquerque - Retina Center, Albuquerque, New Mexico
  - Long Island Vitreoretinal Consultants - Great Neck, Great Neck, New York
  - Vitreoretinal Consultants of NY - Hauppauge, Hauppauge, New York
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Ophthalmic Consultants of the Capital Region - Troy, Troy, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Midwest Retina - Main Office, Dublin, Ohio
  - Retina Northwest - NW Lovejoy, Portland, Oregon
  - Retina Consultants, LLC, Salem, Oregon
  - Mid Atlantic Retina - Philadelphia / Wills Eye Hospital, Bethlehem, Pennsylvania
  - Erie Retinal Research, Erie, Pennsylvania
  - Eye Care Specialists - Kingston, PA, Kingston, Pennsylvania
  - Charleston Neuroscience Institute - Charleston, Charleston, South Carolina
  - Palmetto Retina Center - West Columbia, West Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Charles Retina Specialists - Germantown, Memphis, Tennessee
  - Vanderbilt University Medical School, Nashville, Tennessee
  - Austin Retina Associates - Central, Austin, Texas
  - Texas Retina Associates - Fort Worth, Fort Worth, Texas
  - Medical Center Ophthalmology Associates - Northwest, San Antonio, Texas
  - Retina Consultants of Texas - San Antonio Medical Center, San Antonio, Texas
  - Retina Consultants of Texas (Retina Consultants of Houston) - Texas Medical Center, The Woodlands, Texas
  - Retina Consultants of Texas - The Woodlands, The Woodlands, Texas
  - The University of Vermont Medical Center (Fletcher Allen Health Care) - Main Campus, Burlington, Vermont
  - Spokane Eye Clinical Research, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin
- Argentina (2):
  - Organizacion Medica de Investigacion (OMI), Buenos Aires, Ciudad Auton. de Buenos Aires
  - OFTALMOS, Instituto Oftalmologico de Alta Complejidad, Buenos Aires, Ciudad Auton. de Buenos Aires
- Australia (5):
  - Eyeclinic Albury Wodonga, Albury, New South Wales
  - Marsden Eye Surgery Center, Parramatta, New South Wales
  - Sydney Retina Clinic, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Hobart Eye Surgeons, Hobart, Tasmania
- Austria (5):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt, Carinthia
  - Medizinische Universität Graz, Graz, Styria
  - Kepler Universitätsklinikum Campus III, Linz, Upper Austria
  - Konventhospital Barmherzige Brüder Linz, Linz, Upper Austria
  - Hanusch-Krankenhaus Wien, Vienna
- Bulgaria (6):
  - SEHAT Pentagram, Sofia
  - Spec. Hosp. for Active Treatment for Eye Diseases Zrenie, Sofia
  - University Multiprofile Hospital For Active Treatment 'Alexandrovska' EAD, Sofia
  - Multiprofile Hospital for Active Treatment Sveta Sofia | Internal Diseases Department, Sofia
  - Specialized Hospital For Active Treatment of Eye Diseases Zora, Sofia
  - Sveta Petka Eye Hospital, Varna
- Canada (3):
  - St.Joseph's Health Care-London, London, Ontario
  - Toronto Retina Institute, Toronto, Ontario
  - Institut de l'Oeil des Laurentides, Boisbriand, Quebec
- China (31):
  - The Second Hospital of Anhui medical university, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University (East), Beijing, Dongcheng District
  - The 1st Affiliated Hospital Fujian Medical University, Fuzhou, Fujian
  - Guangzhou Aier Eye Hospital, Guangzhou, Guangdong
  - Hebei eye hospital, Hebei, Hebei
  - Shijiazhuang General Hospital, Shijiazhuang, Hebei
  - Henan Provincial Eye Hospital, Henan, Henan
  - Tongji Hosp. of Tongji Med Coll, Huazhong Uni of Sci & Tech., Wuhan, Hubei
  - Union Hospt Tongji Medical Colleg. Huazhong univ. Scien&Tech, Wuhan, Hubei
  - The First People's Hospital of Xuzhou, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - Eye Center of the second Bethune Hospital, jinlin University, Changchun, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - Shenyang He Eye Specialist Hospital, Shenyang, Liaoning
  - People's Hospital of Ningxia Hui Autonomous Region - Opthalmology, Ningxia, Ningxia
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Aier Eye Hospital (Chengdu), Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The 1st Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - ZheJiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The Affiliated Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Beijing Aier Intech Eye Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Chongqing Aier Ophthalmology Hospital, Chongqing
  - Shanghai Tongji Hospital of Tongji University, Shanghai
  - Shanghai General Hospital, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjin Eye Hospital, Tianjin
  - Tianjin Medical University Eye Hospital, Tianjin
- Czechia (7):
  - Fakultní Nemocnice Hradec Kralové, Hradec Králové
  - Fakultní nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Plzen - Lochotin, Plzen-Lochotin
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Charles University in Prague, Prague
  - Lexum a.s., Evropska ocni klinika, Prague
  - Axon Clinical, s.r.o., Prague
- Estonia (2):
  - AS Ida-Tallinna Keskhaigla - Oftalmoloogiakeskus, Tallinn
  - Sihtasutus Tartu Ülikooli Kliinikum - Silmakliinik, Tartu
- France (3):
  - Centre d'Ophtalmologie - Paradis-Monticelli, Marseille
  - AP-HP - Hopital Lariboisiere, Paris
  - Centre ophtalmologique Saint-Exupéry, Saint-Cyr-sur-Loire
- Georgia (4):
  - LTD "Clinic LJ" - Opthalmology, Kutaisi
  - JSC "Evex Hospitals', Tbilisi
  - LTD "Innova", Tbilisi
  - LTD "Chichua Medical Center MZERA", Tbilisi
- Hungary (2):
  - Budapest Retina Associates, Budapest
  - Szent-Gyorgyi Albert Orvostudomanyi Egyetem, Szeged
- Israel (7):
  - Rambam Health Corporation, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Assuta Medical Centers - HaShalom, Tel Aviv
- Italy (7):
  - Azienda Ospedaliera Policlinico Universitario Tor Vergata, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Fondazione G.B.Bietti Per Lo Studio E La Ricerca In Oftalmologia, Rome, Lazio
  - ASST Fatebenefratelli Sacco, Milan, Lombardy
  - Ospedale San Raffaele s.r.l. - Oculistica, Milan, Lombardy
  - Azienda Ospedaliero-Universitaria Di Cagliari, Cagliari, Sardinia
  - A.O. di Perugia, Perugia, Umbria
- Japan (49):
  - Daiyukai Daiichi Hospital, Ichinomiya, Aichi-ken
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Southern Tohoku Eye Clinic, Kōriyama, Fukushima
  - Gunma University Hospital, Maebashi, Gunma
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - KKR Sapporo Medical Center, Sapporo, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Kozawa Eye Hospital and Diabetes Center, Mito, Ibaraki
  - Kanazawa Medical University Hospital, Kahoku-gun, Ishikawa-ken
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Medical corporation Eiwakai Dannoue Ophthalmology clinic, Kawasaki, Kanagawa
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Otakeganka Tsukimino Clinic, Yamato, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Shinshu University Hospital, Matsumoto, Nagano
  - Nara Medical University Hospital, Kashihara, Nara
  - Oita University Hospital, Yufu, Oita Prefecture
  - Kurashiki Medical Center, Kurashiki, Okayama-ken
  - Okayama University Hospital, Okayama, Okayama-ken
  - University of the Ryukyus Hospital, Nakagami, Okinawa
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kansai Medical University Medical Center, Moriguchi, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - St.Luke's International Hospital, Chuoku, Tokyo
  - Nishikasai Inouye Eye Hospital, Edogawa-ku, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Hachiōji, Tokyo
  - Tokiwadai Muranaka Eye Clinic, Itabashi-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - University of Yamanashi Hospital, Chūō, Yamanashi
  - Akita University Hospital, Akita
  - Hayashi Eye Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Hiroshima University Hospital, Hiroshima
  - University of Miyazaki Hospital, Miyazaki
  - Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Japanese Red Cross Saitama Hospital, Saitama
  - Tokushima University Hospital, Tokushima
  - Japanese Red Cross Wakayama Medical center, Wakayama
  - Yamagata University Hospital, Yamagata
- Latvia (3):
  - Department of Ophthalmology, Riga
  - Latvian American Eye Center, Riga
  - Riga East Clinical University Hospital "Gailezers", Riga
- Lithuania (3):
  - Hospital of LT University of Health Sciences Kaunas Clinics, Kaunas
  - PI Klaipedos University Hospital, Klaipėda
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Portugal (5):
  - ALM Oftalmolaser - Oftalmologia Medica e Cirurgica, Lisbon, Lisbon District
  - AIBILI, Coimbra
  - Espaco Medico de Coimbra, Coimbra
  - Centro Hospitalar Universitario do Porto, Porto
  - Centro Hospitalar Vila Nova de Gaia e Espinho | Unit 1 - Clinical Research Center, Porto
- Russia (2):
  - Scientific Research Institution of Ophthalmic Diseases, Moscow
  - FBSI IRTC Eye Microsurgery n.a. acad. S.N. Fyodorov, Moscow
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - Clinical hospital center Zvezdara, Belgrade
  - Klinicki centar Vojvodine, Novi Sad
- Singapore (2):
  - National University Hospital Medical Centre, Singapore
  - Singapore National Eye Centre, Singapore
- Slovakia (4):
  - Fakultna nemocnica Nitra, Nitra
  - Nemocnica s Poliklinikou Trebisov, Svet zdravia a.s., Trebišov
  - Fakultna nemocnica Trencin, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina, Žilina
- South Korea (7):
  - Nune Eye Hospital - Retina Center Ophthalmology, Seoul, Gangnam-gu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Asan Medical Center - Oncology Department, Seoul, Seoul Teugbyeolsi
  - Pusan National University Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Seoul National University Hospital (b), Seoul
  - Samsung Medical Center - Oncology Department, Seoul
- Spain (7):
  - Instituto Oftalmologico Gomez-Ulla S.L. - Oftalmologia, Santiago de Compostela, A Coruña
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau | Gynecology Department, Barcelona
  - Hospital Universitario Reina Sofia - Oftalmologia, Córdoba
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Y Politecnico La Fe - Oftalmologia, Valencia
  - Hospital Universitario Miguel Servet - Oftalmologia, Zaragoza
- Switzerland (3):
  - RétinElysée, Lausanne, Canton of Vaud
  - Berner Augenklinik am Lindenhofspital, Bern
  - Stadtspital Triemli, Zurich
- Taiwan (3):
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District
- Ukraine (3):
  - Private Enterprise Private Production Company "Acinus", Treatment and Diagnostic Center, Kropyvnytskyi
  - Centralna Polyclinica MVS Ukraiiny, Kyiv
  - Poltava Regional Clinical Hospital n.a. M.V. Skliphosovskyi, Poltava

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Chang A, Sun X, Iida T, Lai TYY, Wong TY, Cheung CMG, Lee WK, Zhang X, Schulze A, Schmidt-Ott UM, Zhao M, Hasanbasic Z, Leal S, Chen SJ; PULSAR study investigators. Intravitreal aflibercept 8 mg versus 2 mg in Asian patients with neovascular age-related macular degeneration: 48-week analysis of the Phase 3 PULSAR trial. Asia Pac J Ophthalmol (Phila). 2026 Jan-Feb;15(1):100278. doi: 10.1016/j.apjo.2026.100278. Epub 2026 Jan 8. PMID 41519383
- [Derived] Lee WK, Wong TY, Chen SJ, Sun X, Cheung CMG, Silva R, Ricci F, Zhang X, Machewitz T, Schulze A, Schmidt-Ott UM, Zhao M, Hasanbasic Z, Leal S, Iida T; PULSAR Study Investigators. Aflibercept 8 mg in Polypoidal Choroidal Vasculopathy: Post Hoc Analysis of the PULSAR Randomized Clinical Trial. JAMA Ophthalmol. 2025 Dec 18. doi: 10.1001/jamaophthalmol.2025.5098. Online ahead of print. PMID 41411005
- [Derived] Korobelnik JF, Lanzetta P, Leal S, Holz FG, Clark WL, Eichenbaum D, Iida T, Sun X, Berliner AJ, Schulze A, Zhao M, Schmelter T, Schmidt-Ott U, Zhang X, Morgan-Warren P, Hasanbasic Z, Vitti R, Chu KW, Reed K, Bhore R, Cheng Y, Bai Z, Hirshberg B, Yancopoulos GD, Wong TY; PULSAR Investigators. Intravitreal Aflibercept 8 mg in Neovascular Age-Related Macular Degeneration: Ninety-Six-Week Results from the Randomized Phase 3 PULSAR Trial. Ophthalmology. 2026 Jan;133(1):39-50. doi: 10.1016/j.ophtha.2025.08.022. Epub 2025 Aug 26. PMID 40876598
- [Derived] Lanzetta P, Korobelnik JF, Heier JS, Leal S, Holz FG, Clark WL, Eichenbaum D, Iida T, Xiaodong S, Berliner AJ, Schulze A, Schmelter T, Schmidt-Ott U, Zhang X, Vitti R, Chu KW, Reed K, Rao R, Bhore R, Cheng Y, Sun W, Hirshberg B, Yancopoulos GD, Wong TY; PULSAR Investigators. Intravitreal aflibercept 8 mg in neovascular age-related macular degeneration (PULSAR): 48-week results from a randomised, double-masked, non-inferiority, phase 3 trial. Lancet. 2024 Mar 23;403(10432):1141-1152. doi: 10.1016/S0140-6736(24)00063-1. Epub 2024 Mar 7. PMID 38461841

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 251 centers in 27 countries/regions with first participant first visit on 20-AUG-2020 and last participant last visit (Week 156) on 07-Aug-2024.
Pre-assignment Details: Overall, 1395 participants were screened, of whom 383 participants did not complete screening, 1 participant was randomized in error although he/she did not complete screening and had withdrawn consent. A total of 1011 participants were randomized in nearly equal numbers to 1 of the 3 treatment groups.
Groups:
- Aflibercept 2q8 (Week 0-96) / HD (up to Week 156): Participants enrolled in main study received aflibercept 2 mg administered every 8 weeks after 3 initial injections at 4-week intervals up to 96 weeks. Participants enrolled in the extension originally assigned to 2q8 in main study and switched to high dose aflibercept starting at Week 96.
- Aflibercep HDq12 (Week 0-156): Participants enrolled in main study received high dose (HD) aflibercept administered every 12 weeks after 3 initial injections at 4-week intervals, up to 96 weeks. Participants enrolled in the extension continued with HD aflibercept at their latest dosing interval at Week 96.
- Aflibercept HDq16 (Week 0-156): Participants enrolled in main study received high dose (HD) aflibercept administered every 16 weeks after 3 initial injections at 4-week intervals, up to 96 weeks. Participants enrolled in the extension continued with HD aflibercept at their latest dosing interval at Week 96.
Period: Main Study
Arm/Group | Aflibercept 2q8 (Week 0-96) / HD (up to Week 156) | Aflibercep HDq12 (Week 0-156) | Aflibercept HDq16 (Week 0-156)
Started (Treated) | 336 | 335 | 338
Completed (Completed study treatment until Week 96) | 286 | 291 | 292
Not Completed | 50 | 44 | 46
Not completed — Adverse Event | 9 | 5 | 8
Not completed — Physician Decision | 3 | 3 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Lost to Follow-up | 3 | 3 | 4
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Withdrawal by Subject | 14 | 20 | 20
Not completed — Death | 10 | 7 | 7
Not completed — COVID-19 pandemic | 2 | 2 | 2
Not completed — Other | 7 | 3 | 2
Period: Extension Phase
Arm/Group | Aflibercept 2q8 (Week 0-96) / HD (up to Week 156) | Aflibercep HDq12 (Week 0-156) | Aflibercept HDq16 (Week 0-156)
Started (Enrolled in extension) | 208 | 210 | 207
Treated | 208 | 210 | 207
Completed (Completed study treatment through Week 156) | 187 | 186 | 191
Not Completed | 21 | 24 | 16
Not completed — Other | 1 | 0 | 0
Not completed — Logistical problems | 0 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Adverse Event | 2 | 3 | 1
Not completed — Death | 4 | 7 | 2
Not completed — Withdrawal by Subject | 11 | 11 | 7

BASELINE CHARACTERISTICS:
Population: Full analysis set: included all participants who had been randomly assigned to study treatment and who received at least 1 dose of study treatment.
Groups:
- Aflibercept 2q8: Participants received aflibercept 2 mg administered every 8 weeks after 3 initial injections at 4-week intervals, up to 96 weeks.
- Aflibercept HDq12: Participants received high dose (HD) aflibercept administered every 12 weeks after 3 initial injections at 4-week intervals, up to 96 weeks. Participants in this group can have their treatment intervals adjusted according to pre-specified dose regimen modification (DRM) criteria
- Aflibercept HDq16: Participants received high dose (HD) aflibercept administered every 16 weeks after 3 initial injections at 4-week intervals, up to 96 weeks. Participants in this group can have their treatment intervals adjusted according to pre-specified DRM criteria
- Total: Total of all reporting groups
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16 | Total
Number analyzed (Participants) | 336 | 335 | 338 | 1009
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.2 (8.8) | 74.7 (7.9) | 74.5 (8.5) | 74.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 182 | 180 | 550
  Male | 148 | 153 | 158 | 459
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 9 | 28
  Not Hispanic or Latino | 322 | 322 | 326 | 970
  Unknown or Not Reported | 2 | 6 | 3 | 11
Baseline BCVA measured by the ETDRS letter score [Mean (Standard Deviation); unit: scores on a scale] — Visual function of the study eye was assessed at a distance of 4 meters using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. BCVA scale range is 0 (worst) to 100 (best).
  scores on a scale | 58.9 (14.0) | 59.9 (13.4) | 60.0 (12.4) | 59.6 (13.3)
Baseline choroidal neovascularization (CNV) size [Mean (Standard Deviation); unit: mm²] — Population: Full analysis set, except 1 participant who did not have a valid baseline measure.
  mm²
    number analyzed (Participants) | 336 | 335 | 337 | 1008
    (all) | 6.3593 (5.0394) | 5.9768 (4.8306) | 6.5459 (5.5315) | 6.2946 (5.1433)
Baseline total lesion area [Mean (Standard Deviation); unit: mm²] — Population: Full analysis set, except 2 participants who did not have a valid baseline measure.
  mm²
    number analyzed (Participants) | 336 | 335 | 336 | 1007
    (all) | 6.8647 (5.4145) | 6.3820 (5.0664) | 6.8814 (5.6514) | 6.7097 (5.3827)
Baseline central subfield retinal thickness (CST) [Mean (Standard Deviation); unit: µm] — Population: Full analysis set, except 3 participants who did not have a valid baseline measure.
  µm
    number analyzed (Participants) | 335 | 335 | 336 | 1006
    (all) | 367.1 (133.6) | 370.3 (123.7) | 370.7 (132.7) | 369.3 (130.0)
Baseline NEI-VFQ-25 total score [Mean (Standard Deviation); unit: scores on a scale] — NEI-VFQ-25 = National Eye Institute Visual Functioning Questionnaire-25
  NEI VFQ-25 was a 25-item questionnaire that gave a score on a scale from 0 (worst) to 100 (best = no vision problems) Population: Full analysis set, with the participants who completed the NEI-VFQ-25 at baseline.
  scores on a scale
    number analyzed (Participants) | 317 | 321 | 316 | 954
    (all) | 77.8082 (14.4206) | 76.3575 (15.1213) | 77.6670 (15.3980) | 77.2733 (14.9843)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in BCVA Measured by the ETDRS Letter Score at Week 48
Description: Visual function of the study eye was assessed at a distance of 4 meters using the ETDRS BCVA letter score. BCVA scale range is 0 (worst) to 100 (best).
Time Frame: At baseline and Week 48
Population: Full analysis set: included all participants who had been randomly assigned to study treatment and who received at least 1 dose of study treatment. Estimand mainly based on hypothetical strategy.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16
Number analyzed (Participants) | 336 | 335 | 338
scores on a scale | 7.03 (0.74) | 6.06 (0.77) | 5.89 (0.72)
Statistical Analysis 1: Comparison: Aflibercept 2q8 vs Aflibercept HDq12; HDq12 - 2q8; Test type: Non-Inferiority — One-sided test (alpha=0.025) for non-inferiority at a 4-letter margin; p = 0.0009, Mixed Models Analysis — Strictly hierarchical testing procedure: Since p-value below significance level 0.025, fixed sequence testing continued with next primary endpoint (HDq16-2q8) / within EMA/PMDA specific hierarchy with secondary endpoint (BCVA at W60, HDq12-2q8); Adjusted for baseline BCVA and randomization strata; Difference in LS means = -0.97, 95% CI 2-sided [-2.87 to 0.92] — Estimation mainly based on hypothetical strategy, i.e. observed data beyond intercurrent events (premature discontinuation of treatment, missing injection, prohibited medication) were censored. Missing/censored data was handled implicitly by MMRM
Statistical Analysis 2: Comparison: Aflibercept 2q8 vs Aflibercept HDq16; HDq16 - 2q8; Test type: Non-Inferiority — One-sided test (alpha=0.025) for non-inferiority at a 4-letter margin; p = 0.0011, Mixed Models Analysis — Strictly hierarchical testing procedure: Since p-value below significance level 0.025, fixed sequence testing continued with secondary endpoint (no IRF no SRF at W16)/within EMA/PMDA specific hierarchy with secondary endpoint (BCVA at W60, HDq16-2q8); Adjusted for baseline BCVA and randomization strata; Difference in LS means = -1.14, 95% CI 2-sided [-2.97 to 0.69] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in BCVA Measured by the ETDRS Letter Score at Week 60
Description: as for outcome 1
Time Frame: At baseline and Week 60
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16
Number analyzed (Participants) | 336 | 335 | 338
scores on a scale | 7.23 (0.68) | 6.37 (0.74) | 6.31 (0.66)
Statistical Analysis 1: Comparison: Aflibercept 2q8 vs Aflibercept HDq12; HDq12 - 2q8; Test type: Non-Inferiority — One-sided test (alpha=0.025) for non-inferiority at a 4-letter margin; p = 0.0002, Mixed Models Analysis — EMA/PMDA specific hierarchy: i.e. secondary endpoint was tested for EMA/PMDA after primary endpoint (HDq12-2q8). Since p-value below significance level 0.025, EMA/PMDA specific fixed sequence testing continued with next primary endpoint (HDq16-2q8); Adjusted for baseline BCVA and randomization strata; Difference in LS means = -0.86, 95% CI 2-sided [-2.57 to 0.84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Aflibercept 2q8 vs Aflibercept HDq16; HDq16 - 2q8; Test type: Non-Inferiority — One-sided test (alpha=0.025) for non-inferiority at a 4-letter margin; p < 0.0001, Mixed Models Analysis — EMA/PMDA specific hierarchy: i.e. secondary endpoint was tested after primary endpoint (HDq16-2q8). Since p-value below significance level 0.025, EMA/PMDA specific fixed sequence testing continued with secondary endpoint test (no IRF no SRF at W16); Adjusted for baseline BCVA and randomization strata; Difference in LS means = -0.92, 95% CI 2-sided [-2.51 to 0.66] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With no Intraretinal Fluid (IRF) and no Subretinal Fluid (SRF) in Central Subfield at Week 16
Time Frame: At Week 16
Population: Full analysis set: included all participants who had been randomly assigned to study treatment and who received at least 1 dose of study treatment. Estimand mainly based on hypothetical strategy.
  The Overall Number of Participants Analyzed is not consistent with numbers provided in the Overall Number of Baseline Participants due to missing assessment at the respective visit. These participants with missing assessments were not included in the analysis.
Measure: Number; unit: Percentage of participants
Groups:
- All Aflibercept HD: Included all participants from aflibercept HDq12 and aflibercept HDq16
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16 | All Aflibercept HD
Number analyzed (Participants) | 335 | 333 | 334 | 667
Percentage of participants | 51.6 | 61.6 | 65.0 | 63.3
Statistical Analysis 1: Comparison: Aflibercept 2q8 vs All Aflibercept HD; All HD - 2q8; Test type: Superiority — One sided test (alpha = 0.025) for superiority; p = 0.0002, Cochran-Mantel-Haenszel — Strictly hierarchical testing procedure to adjust for multiplicity; CMH test stratified by baseline BCVA and randomization strata; Difference = 11.733, 95% CI 2-sided [5.263 to 18.204] — Estimation mainly based on hypothetical strategy, i.e. observed data beyond intercurrent events (premature discontinuation of treatment, missing injection, prohibited medication) were censored. Missing/censored data was imputed by LOCF approach

4. Secondary Outcome: Percentage of Participants Gaining at Least 15 Letters in BCVA From Baseline at Week 48
Time Frame: At baseline and Week 48
Population: Full analysis set: included all participants who had been randomly assigned to study treatment and who received at least 1 dose of study treatment.
  The Overall Number of Participants Analyzed is not consistent with numbers provided in the Overall Number of Baseline Participants due to 1 participant per each treatment group with no post-baseline BCVA. These participants with missing assessments were not included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16
Number analyzed (Participants) | 335 | 334 | 337
Percentage of participants | 22.1 | 20.7 | 21.7
Statistical Analysis 1: Comparison: Aflibercept 2q8 vs Aflibercept HDq12; HDq12 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.5704, Cochran-Mantel-Haenszel — Nominal p-value, not adjusted for multiplicity; CMH test stratified by baseline BCVA and randomization strata; Difference = -1.748, 95% CI 2-sided [-7.784 to 4.287] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Aflibercept 2q8 vs Aflibercept HDq16; HDq16 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.7611, Cochran-Mantel-Haenszel — Nominal p-value, not adjusted for multiplicity; CMH test stratified by baseline BCVA and randomization strata; Difference = -0.939, 95% CI 2-sided [-6.997 to 5.119] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Percentage of Participants Achieving an ETDRS Letter Score of at Least 69 (Approximate 20/40 Snellen Equivalent) at Week 48
Time Frame: At Week 48
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16
Number analyzed (Participants) | 335 | 334 | 337
Percentage of participants | 57.9 | 56.9 | 54.3
Statistical Analysis 1: Comparison: Aflibercept 2q8 vs Aflibercept HDq12; HDq12 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.9554, Cochran-Mantel-Haenszel — Nominal p-value, not adjusted for multiplicity; CMH test stratified by baseline BCVA and randomization strata; Difference = -0.182, 95% CI 2-sided [-6.565 to 6.200] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Aflibercept 2q8 vs Aflibercept HDq16; HDq16 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.4834, Cochran-Mantel-Haenszel — Nominal p-value, not adjusted for multiplicity; CMH test stratified by baseline BCVA and randomization strata; Difference = -2.221, 95% CI 2-sided [-8.435 to 3.994] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Change in Choroidal Neovascularization (CNV) Size From Baseline to Week 48
Time Frame: At baseline and Week 48
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16
Number analyzed (Participants) | 336 | 335 | 338
mm^2 | -2.43 (0.31) | -3.65 (0.28) | -2.91 (0.29)
Statistical Analysis 1: Comparison: Aflibercept 2q8 vs Aflibercept HDq12; HDq12 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.0009, Mixed Models Analysis — Nominal p-value, not adjusted for multiplicity; Adjusted for baseline CNV size and randomization strata; Difference in LS means = -1.22, 95% CI 2-sided [-1.94 to -0.51] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Aflibercept 2q8 vs Aflibercept HDq16; HDq16 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.2076, Mixed Models Analysis — Nominal p-value, not adjusted for multiplicity; Adjusted for baseline CNV size and randomization strata; Difference in LS means = -0.48, 95% CI 2-sided [-1.22 to 0.27] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change in Total Lesion Area From Baseline to Week 48
Time Frame: At baseline and Week 48
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16
Number analyzed (Participants) | 336 | 335 | 338
mm^2 | 0.09 (0.22) | -0.46 (0.19) | -0.35 (0.20)
Statistical Analysis 1: Comparison: Aflibercept 2q8 vs Aflibercept HDq12; HDq12 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.0287, Mixed Models Analysis — Nominal p-value, not adjusted for multiplicity; Adjusted for baseline total lesion area and randomization strata; Difference in LS means = -0.55, 95% CI 2-sided [-1.04 to -0.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Aflibercept 2q8 vs Aflibercept HDq16; HDq16 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.0870, Mixed Models Analysis — Nominal p-value, not adjusted for multiplicity; Adjusted for baseline total lesion area and randomization strata; Difference in LS means = -0.44, 95% CI 2-sided [-0.94 to 0.06] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Percentage of Participants With no Intraretinal Fluid (IRF) and no Subretinal Fluid (SRF) in the Center Subfield at Week 48
Time Frame: At Week 48
Population: Full analysis set: included all participants who had been randomly assigned to study treatment and who received at least 1 dose of study treatment.
  The Overall Number of Participants Analyzed is not consistent with numbers provided in the Overall Number of Baseline Participants due to missing assessments at the respective visit. These participants with missing assessments were not included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16
Number analyzed (Participants) | 335 | 332 | 334
Percentage of participants | 59.4 | 71.1 | 66.8
Statistical Analysis 1: Comparison: Aflibercept 2q8 vs Aflibercept HDq12; HDq12 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.0015, Cochran-Mantel-Haenszel — Nominal p-value, not adjusted for multiplicity; CMH test stratified by baseline BCVA and randomization strata; Difference = 11.725, 95% CI 2-sided [4.527 to 18.923] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Aflibercept 2q8 vs Aflibercept HDq16; HDq16 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.0458, Cochran-Mantel-Haenszel — Nominal p-value, not adjusted for multiplicity; CMH test stratified by baseline BCVA and randomization strata; Difference = 7.451, 95% CI 2-sided [0.142 to 14.760] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Change From Baseline in Central Subfield Retinal Thickness (CST) at Week 48
Time Frame: At baseline and Week 48
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: µm
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16
Number analyzed (Participants) | 336 | 335 | 338
µm | -136.25 (4.24) | -147.37 (4.01) | -146.76 (3.76)
Statistical Analysis 1: Comparison: Aflibercept 2q8 vs Aflibercept HDq12; HDq12 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.0283, Mixed Models Analysis — Nominal p-value, not adjusted for multiplicity; Adjusted for baseline CST and randomization strata; Difference in LS means = -11.12, 95% CI 2-sided [-21.06 to -1.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Aflibercept 2q8 vs Aflibercept HDq16; HDq16 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.0321, Mixed Models Analysis — Nominal p-value, not adjusted for multiplicity; Adjusted for baseline CST and randomization strata; Difference in LS means = -10.51, 95% CI 2-sided [-20.12 to -0.90] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change From Baseline in National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ-25) Total Score at Week 48
Description: NEI VFQ-25 was a 25-item questionnaire that gave a score on a scale from 0 (worst) to 100 (best = no vision problems)
Time Frame: At baseline and Week 48
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16
Number analyzed (Participants) | 336 | 335 | 338
scores on a scale | 4.22 (0.70) | 3.50 (0.70) | 3.35 (0.72)
Statistical Analysis 1: Comparison: Aflibercept 2q8 vs Aflibercept HDq12; HDq12 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.3817, Mixed Models Analysis — Nominal p-value, not adjusted for multiplicity; Adjusted for baseline NEI-VFQ-25 total score and randomization strata; Difference in LS means = -0.72, 95% CI 2-sided [-2.35 to 0.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Aflibercept 2q8 vs Aflibercept HDq16; HDq16 - 2q8; Test type: Equivalence — Two sided test (alpha = 0.05); p = 0.3070, Mixed Models Analysis — Nominal p-value, not adjusted for multiplicity; Adjusted for baseline NEI-VFQ-25 total score and randomization strata; Difference in LS means = -0.87, 95% CI 2-sided [-2.55 to 0.80] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Systemic Exposure to Aflibercept as Assessed by Plasma Concentrations of Free, Adjusted Bound and Total Aflibercept From Baseline Through Week 48
Time Frame: Up to Week 48
Population: Pharmacokinetic analysis set: included all participants who received any study treatment and who had at least 1 non-missing drug concentration measurement following the first dose of study treatment
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16
Number analyzed (Participants) | 308 | 313 | 313
mg/L
  Week 4: number analyzed (Participants) | 287 | 295 | 299
  Week 4 | NA (NA) — Not calculated (less than 2/3 of values per timepoint are >= Lower level of quantification (LLOQ) for geometric mean calculation). | NA (NA) — Not calculated (less than 2/3 of values per timepoint are >= Lower level of quantification (LLOQ) for geometric mean calculation). | NA (NA) — Not calculated (less than 2/3 of values per timepoint are >= Lower level of quantification (LLOQ) for geometric mean calculation).
  Visit 5: within 3 to 7 days after the Week 8: number analyzed (Participants) | 263 | 269 | 255
  Visit 5: within 3 to 7 days after the Week 8 | 0.03 (70.29) | 0.14 (78.69) | 0.13 (82.50)
  Week 12: number analyzed (Participants) | 292 | 291 | 302
  Week 12 | NA (NA) — Not calculated (less than 2/3 of values per timepoint are >= Lower level of quantification (LLOQ) for geometric mean calculation). | 0.02 (81.35) | 0.02 (84.06)
  Week 28: number analyzed (Participants) | 268 | 291 | 283
  Week 28 | NA (NA) — Not calculated (less than 2/3 of values per timepoint are >= Lower level of quantification (LLOQ) for geometric mean calculation). | NA (NA) — Not calculated (less than 2/3 of values per timepoint are >= Lower level of quantification (LLOQ) for geometric mean calculation). | NA (NA) — Not calculated (less than 2/3 of values per timepoint are >= Lower level of quantification (LLOQ) for geometric mean calculation).
  Week 48: number analyzed (Participants) | 265 | 275 | 273
  Week 48 | NA (NA) — Not calculated (less than 2/3 of values per timepoint are >= Lower level of quantification (LLOQ) for geometric mean calculation). | NA (NA) — Not calculated (less than 2/3 of values per timepoint are >= Lower level of quantification (LLOQ) for geometric mean calculation). | NA (NA) — Not calculated (less than 2/3 of values per timepoint are >= Lower level of quantification (LLOQ) for geometric mean calculation).

12. Secondary Outcome: Incidence of Treatment-emergent Anti-drug Antibodies (ADA) Response
Time Frame: Up to week 96
Measure: Count of Participants; unit: Participants
Groups:
- All Aflibercept HD: All participants from aflibercept HDq12 (Week 0-96) and aflibercept HDq16 (Week 0-96).
Arm/Group | Aflibercept 2q8 | Aflibercept HDq12 | Aflibercept HDq16 | All Aflibercept HD
Number analyzed (Participants) | 284 | 295 | 295 | 590
Participants
  Treatment-emergent positive or Treatment-boosted, maximum ADA titers - Low (< 1000) | 8 | 14 | 13 | 27
  Treatment-emergent positive or Treatment-boosted, maximum ADA titers - Moderate (1000-10000) | 0 | 0 | 0 | 0
  Treatment-emergent positive or Treatment-boosted, maximum ADA titers - High (> 10000) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through Week 96, from first dosing up to 30 days after last dosing (active or sham procedure). Through Week 156, from first dosing up to 30 days after last dosing (active or sham procedure) or the Week 156 visit, whichever was later. AE reporting for all-cause mortality considers all deaths occurred at any time during the study before the last contact.
Description: Ocular TEAEs in study eye and non-ocular TEAEs (ocular TEAEs in fellow eye are excluded)
Groups:
- Aflibercept 2q8 (Week 0- 96): Participants enrolled in main study received aflibercept 2 mg administered every 8 weeks after 3 initial injections at 4-week intervals.
- Aflibercept HDq12 (Week 0- 96): Participants enrolled in main study received high dose (HD) aflibercept administered every 12 weeks after 3 initial injections at 4-week intervals. Participants in this group could have their treatment intervals adjusted according to pre-specified dose regimen modification (DRM) criteria.
- Aflibercept HDq16 (Week 0- 96): Participants enrolled in main study received high dose (HD) aflibercept administered every 16 weeks after 3 initial injections at 4-week intervals. Participants in this group could have their treatment intervals adjusted according to pre-specified dose regimen modification (DRM) criteria.
- All Aflibercept HD (Week 0- 96): All participants from aflibercept HDq12 (Week 0-96) and aflibercept HDq16 (Week 0-96).
- Aflibercept 2q8/HD (Week 0- 156): Participants enrolled in the extension originally assigned to 2q8 in main study and switched to high dose aflibercept every 12 weeks starting at Week 96. Participants in this group could have their treatment intervals adjusted in the extension according to pre-specified dose regimen modification (E-DRM) criteria.
- Aflibercept HDq12 (Week 0- 156): Participants enrolled in the extension originally assigned to HDq12 in main study and continued with HD aflibercept at their latest dosing interval at Week 96. Participants in this group could have their treatment intervals adjusted in the extension according to pre-specified dose regimen modification (E-DRM) criteria.
- Aflibercept HDq16 (Week 0- 156): Participants enrolled in the extension originally assigned to HDq16 in main study and continued with HD aflibercept at their latest dosing interval at Week 96. Participants in this group could have their treatment intervals adjusted in the extension according to pre-specified dose regimen modification (E-DRM) criteria.
- All Aflibercept HD (Week 0- 156): All participants from aflibercept HDq12 (Week 0-156) and aflibercept HDq16 (Week 0-156). Participants in this group could have their treatment intervals adjusted in the extension according to pre-specified dose regimen modification (E-DRM) criteria.
Arm/Group | Aflibercept 2q8 (Week 0- 96) | Aflibercept HDq12 (Week 0- 96) | Aflibercept HDq16 (Week 0- 96) | All Aflibercept HD (Week 0- 96) | Aflibercept 2q8/HD (Week 0- 156) | Aflibercept HDq12 (Week 0- 156) | Aflibercept HDq16 (Week 0- 156) | All Aflibercept HD (Week 0- 156)
All-Cause Mortality (participants affected / at risk) | 12/336 | 11/335 | 7/338 | 18/673 | 4/208 | 7/210 | 2/207 | 9/417
Serious Adverse Events (participants affected / at risk) | 69/336 | 83/335 | 72/338 | 155/673 | 49/208 | 61/210 | 61/207 | 122/417
Other Adverse Events (participants affected / at risk) | 179/336 | 163/335 | 180/338 | 343/673 | 136/208 | 120/210 | 135/207 | 255/417
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2q8 (Week 0- 96) (N=336) | Aflibercept HDq12 (Week 0- 96) (N=335) | Aflibercept HDq16 (Week 0- 96) (N=338) | All Aflibercept HD (Week 0- 96) (N=673) | Aflibercept 2q8/HD (Week 0- 156) (N=208) | Aflibercept HDq12 (Week 0- 156) (N=210) | Aflibercept HDq16 (Week 0- 156) (N=207) | All Aflibercept HD (Week 0- 156) (N=417)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (3) | 2 (2) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 3 (3) | 5 (5) | 8 (8)
Dry age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Macular detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 2 (2) | 3 (3) | 5 (5) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Retinal haemorrhage (Eye disorders) | 1 (6) | 2 (2) | 2 (2) | 4 (4) | 1 (6) | 1 (1) | 2 (2) | 3 (3)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Haemorrhagic cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic vascular thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 5 (5) | 5 (5) | 10 (10) | 2 (2) | 3 (3) | 3 (3) | 6 (6)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Q fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Systemic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 3 (3) | 4 (5) | 1 (1) | 1 (1) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (3) | 1 (1) | 1 (1) | 2 (4) | 3 (5)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 3 (4) | 8 (9) | 2 (2) | 4 (4) | 3 (4) | 7 (8)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff tear arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oesophageal carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Carotid aneurysm rupture (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial mass (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stroke in evolution (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bladder stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough variant asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 1 (2) | 3 (3) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 5 (5)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disability (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Artificial urinary sphincter implant (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Giant cell arteritis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2q8 (Week 0- 96) (N=336) | Aflibercept HDq12 (Week 0- 96) (N=335) | Aflibercept HDq16 (Week 0- 96) (N=338) | All Aflibercept HD (Week 0- 96) (N=673) | Aflibercept 2q8/HD (Week 0- 156) (N=208) | Aflibercept HDq12 (Week 0- 156) (N=210) | Aflibercept HDq16 (Week 0- 156) (N=207) | All Aflibercept HD (Week 0- 156) (N=417)
Cataract (Eye disorders) | 22 (22) | 29 (29) | 32 (33) | 61 (62) | 27 (29) | 34 (37) | 33 (35) | 67 (72)
Retinal haemorrhage (Eye disorders) | 19 (21) | 16 (16) | 17 (20) | 33 (36) | 17 (22) | 11 (11) | 11 (15) | 22 (26)
Visual acuity reduced (Eye disorders) | 24 (31) | 21 (24) | 23 (34) | 44 (58) | 16 (23) | 15 (17) | 14 (16) | 29 (33)
Vitreous floaters (Eye disorders) | 16 (17) | 5 (6) | 17 (19) | 22 (25) | 12 (13) | 2 (2) | 18 (20) | 20 (22)
Bronchitis (Infections and infestations) | 10 (11) | 8 (8) | 4 (4) | 12 (12) | 11 (11) | 7 (8) | 6 (7) | 13 (15)
COVID-19 (Infections and infestations) | 60 (64) | 58 (59) | 70 (73) | 128 (132) | 50 (59) | 44 (45) | 59 (62) | 103 (107)
Nasopharyngitis (Infections and infestations) | 30 (40) | 18 (25) | 27 (31) | 45 (56) | 28 (46) | 20 (33) | 28 (38) | 48 (71)
Urinary tract infection (Infections and infestations) | 18 (20) | 12 (12) | 14 (19) | 26 (31) | 17 (20) | 11 (11) | 14 (20) | 25 (31)
Intraocular pressure increased (Investigations) | 10 (19) | 12 (20) | 11 (20) | 23 (40) | 8 (20) | 12 (21) | 8 (12) | 20 (33)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 12 (13) | 11 (12) | 23 (25) | 7 (9) | 6 (7) | 14 (15) | 20 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (31) | 17 (27) | 14 (15) | 31 (42) | 14 (24) | 11 (24) | 14 (15) | 25 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 8 (8) | 13 (14) | 21 (22) | 15 (22) | 6 (6) | 12 (16) | 18 (22)
Hypertension (Vascular disorders) | 18 (21) | 22 (26) | 23 (23) | 45 (49) | 18 (20) | 21 (25) | 15 (15) | 36 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT04423718/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04423718/SAP_001.pdf